CLINICAL TRIAL: NCT05382923
Title: Circadian Acclimatization of Performance, Sleep, and 6-sulphatoxymelatonin Using Multiple Phase-Shifting Stimuli
Brief Title: Facilitating Adjustment to Simulated Jet Lag
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Arizona (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Shawn Youngstedt, Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2011240758
Record Dates: First submitted 2022-03-02; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Circadian Rhythm Sleep Disorder, Jet Lag Type
MeSH Terms: conditions — Jet Lag Syndrome | interventions — Exercise; Melatonin

STUDY DESIGN:
Intervention Model Description: Random assignment to one of three conditions
Who Masked: Participant
Masking Description: Participants are informed that we are exploring different types of stimuli (including exercise, melatonin, and light) to help adjust to simulated jet lag.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bright Light Alone (Experimental): Bright light administered with Re-Timer glasses for 1 hour on 3 consecutive days. Following the 8 hour delay of the light/dark and sleep/wake cycle in the laboratory, the light will be administered, on average at 5:30-6:30 pm, 7:00-8:00 pm, and 9:30-10:30 pm, respectively on these three days.
  Interventions: Behavioral: Bright Light
- Bright Light + Exercise + Melatonin (Experimental): Bright light will be administered with Re-Timer glasses for 1 hour on 3 consecutive days. Following the 8 hour delay of the light/dark and sleep/wake cycle in the laboratory, the light will be administered, on average at 5:30-6:30 pm, 7:00-8:00 pm, and 9:30-10:30 pm, respectively on these three days. Exercise (1 hour at 65-75% heart rate reserve) will be administered on 3 consecutive, at 1:30-2:30 pm, 4:00-5:00 pm, and 6:30-7:30 pm on these days. Melatonin (0.5 mg) will be administered at 6 am, 8:30 am, and 11:00, on the 3 days.
  Interventions: Behavioral: Bright Light + Exercise + Melatonin
- Placebo Control (Placebo Comparator): Dim red light will be administered with Re-Timer glasses for 1 hour on 3 consecutive days. Following the 8 hour delay of the light/dark and sleep/wake cycle in the laboratory, the light will be administered, on average at 5:30-6:30 pm, 7:00-8:00 pm, and 9:30-10:30 pm, respectively on these three days. Placebo tablets (0.5 mg) will be administered at 6 am, 8:30 am, and 11:00, on the 3 days.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Bright Light — 3 consecutive days of 1 hour bright light
  Other Names: Bright Light Treatment
  Arms: Bright Light Alone
Behavioral: Bright Light + Exercise + Melatonin — 3 consecutive days of bright light, exercise, and melatonin
  Other Names: Bright Light Treatment + Treadmill Exercise + Melatonin
  Arms: Bright Light + Exercise + Melatonin
Behavioral: Control — 3 consecutive days of dim red light + light stretching + placbo
  Other Names: Placebo Control
  Arms: Placebo Control

SUMMARY:
The aims of this study are to compare 3 different treatments for circadian adjustment to a laboratory protocol which will mimic westward air travel across 8 time zones. One treatment will involve simply following the new schedule for 3 days. Another treatment will also involve exposure to bright light for 1 hour per day. A third treatment will involve exposure to bright light + exercise for 1 hour per day + consuming a melatonin tablet. Adjustment to the shifted schedule will be assessed by comparing measures of sleep, mood, mental performance, physical performance, and timing of melatonin across the 3 treatment conditions.

DETAILED DESCRIPTION:
Design Overview. Following a 1 week home baseline, N=36 young adults will spend 6 days in the laboratory (Figure 3 and Table 1). Following am 8 h baseline polysomnographic recording (PSG) on Night 1, participants will undergo a 26 h baseline circadian assessment via an ultrashort sleep-wake protocol involving 2 h wake intervals and 1 h sleep intervals, repeated throughout the protocol. Following baseline circadian assessment, participants will be placed on a 16 h wake-8 h sleep schedule in which the wake-sleep and light-dark schedule is delayed 8 h for 3 days (analogous to traveling 8 time zones west). Participants will be randomized to one of 3 treatments (n=12 per treatment) administered each of the 3 days of the shifted schedule: (1) placebo control, (2) bright light, and (3) bright light + exercise + melatonin. PSG recording will occur on the last night of the shifted schedule, followed by an end-of-study 26 h ultrashort sleep wake schedule. On baseline Day 1 and Days 2-3 of the shifted schedule, sleepiness, mood, and mental performance will be assessed every 3 h during wake. During all four 8 h sleep periods, sleep will also be recorded with the Z-machine, which assesses sleep stages from 3 EEG electrodes. During the ultrashort sleep-wake schedules, mental performance, physiological performance, urinary aMT6s, mood, and sleepiness will be measured around-the-clock.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-45 years
2. At least moderate level of habitual physical activity (twice per week, 20 min of aerobic exercise at 60% of maximal effort or higher

Exclusion Criteria:

(1)Having more than one risk factor for coronary artery disease: (2) having any symptom or sign of cardiopulmonary disease; (3) recent shift-work experience (previous 2 months) or travel across multiple time zones (previous 4 weeks); (4) having an abnormal sleep-wake schedule (i.e., reported bedtime before 9:00 pm or after 2:00 am; wake time before 5:00 am or after 10:00 am); (5) being an extreme night owl or morning lark, as assessed by the Horne-Ostberg Mornngness-Eveningness Scale;70 (6) having a high risk sleep apnea or another sleep disorder; (7) depressed mood [Center for Epidemiologic Studies-Depression Scale (CES-D) > 16];71 (7) use of medications likely to distort melatonin excretion or cardiovascular responses to exercise; (8) use of sleeping pills more than 1 night per week; (9) having high sensitivity to light; (10) abuse of alcohol or drugs (amount per week; related problems such as missing work); (11) any physical or mental health condition that would contraindicate participation in exercise or other rigors of the experiment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-07-10 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Change (shift) in the acrophase of urinary 6-sulphatoxymelatonin (aMT6s) excretion | 6.5 days
  Change (shift) in the cosine fitted peak for the assessments (every 90 min) during lab days 2-3 compared with the assessments taken during days 6-7
Change (shift) in the acrophase of the rhythm of the median reaction time | 6.5 days
  Change (shift) in the cosine fitted peak for the assessments (psychomotor vigilance, every 3 h) taken during days 2-3 compared with the assessments taken during days 6-7
Change in sleep duration | 5 days
  Change in total sleep time assessed during night one in the lab and night 5 in the lab duration

SECONDARY OUTCOMES:
Change (shift) in the acrophase of the Total Mood Disturbance composite scale of on the Profile of Mood States questionnaire | 5 days
  Change (shift) in the cosine-fitted peak of the rhythm of total mood disturbance assessed during days 2-3 compared with total mood disturbance assessed during days 6-7
Change (shift) in the acrophase of the Stanford Sleepiness Scale | 5 days
  Change (shift) in the cosine-fitted peak of the rhythm of the Stanford Sleepiness Scale assessed during days 2-3 compared with the Stanford Sleepiness Scale mood disturbance assessed during days 6-7
Change (shift) in the acrophase of the Wingate Anaerobic Performance Test | 5 days
  Change (shift) in the cosine-fitted peak of the rhythm of the Wingate Anaerobic Performance Test assessed on days 2-3 and day 6-7.
Change in sleep recorded with z-machine | 5 days
  Z machine recorded sleep with electrodes on the mastoid bones. Change in sleep assessed in eight 1-h sleep intervals on days 2-3 and days 6-7

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Youngstedt, PhD, Principal Investigator — Univ Arizona; Salma Patel, MD, Principal Investigator — University of Arizona
Locations (1):
- Center Sleep and Circadian Sciences, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
None. We will only share mean data which are de-identified